CLINICAL TRIAL: NCT01952756
Title: Cilostazol Enhances the Number and Functions of Circulating Endothelial Progenitor Cells and Collateral Formation Assessed by Dual-energy 128-row CT Angiography Mediated Through Multiple Mechanisms in Patients With Mild-to-moderate PAOD
Brief Title: Effect of Cilostazol Endothelial Progenitor Cells and Collateral Formation in Peripheral Occlusive Artery Disease (PAOD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCKUH-10103043/BR-100-134
Record Dates: First submitted 2013-09-21; First posted 2013-09-30 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Peripheral Arterial Diseases
Keywords: cilostazol; endothelial progenitor cells; vasculogenesis; angiogenesis; peripheral arterial disease; biomarkers
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Active Comparator): One tablet (100 mg) twice per day for 12 weeks
  Interventions: Drug: Cilostazol
- Dummy Placebo (Placebo Comparator): One tablet twice per day for 12 weeks
  Interventions: Drug: Dummy Placebo

INTERVENTIONS:
Drug: Cilostazol — One tablet (100 mg) twice per day for 12 weeks
  Other Names: Pletaal (brand name)
  Arms: Cilostazol
Drug: Dummy Placebo — One tablet twice per day for 12 weeks
  Other Names: Placebo; Control
  Arms: Dummy Placebo

SUMMARY:
1. The number and function of circulating endothelial progenitor cells (EPCs) are inversely associated with coronary risk factors and atherosclerotic diseases such as PAOD.
2. This double-blind, randomized, placebo-controlled trial to evaluate the effects of cilostazol on human early EPCs and angiogenesis as well as the potential mechanisms of action in patients with mild-to-moderate PAOD.

DETAILED DESCRIPTION:
1. titration of drugs

   1. run-in period: eligible subjects are screened and baseline blood samples are obtained
   2. study period: 12 weeks

      * 24 subjects with cilostazol and 20 subjects with dummy placebo
      * On the first day after the end of the study period, the follow-up data are obtained by the same procedure
   3. blood sampling and measurement of serum biomarkers

      * obtained from peripheral veins in all study subjects at the run-in period and the end of the treatment period of the study
      * sent for isolation, cell culture, and assays of human EPCs
      * also stored for enzyme-linked immunosorbent assay (Stromal cell derived factor-alfa1, adiponectin, soluble thrombomodulin, vascular endothelial growth factor)
2. assays of human EPCs

   1. colony formation by EPCs
   2. quantification of EPCs and apoptotic endothelial cells
   3. chemotactic motility, proliferation/viability and apoptosis assays
3. collateral vessels formation and distal run-off assessed by dual-energy multi-slice computed tomography angiography
4. echocardiographic examinations to evaluate left ventricular functions

ELIGIBILITY:
Inclusion Criteria:

* ankle-brachial index (ABI) less than 0.9 in one or both legs but no obvious symptoms of intermittent claudication

Exclusion Criteria:

* obvious symptoms of intermittent claudication
* severe PAD (Fontaine grading > 3) or critical limb ischemia in at least one leg
* severe liver dysfunction (transaminases >10 times of upper normal limit, history of liver cirrhosis, or hepatoma)
* > stage 4 chronic kidney disease (end-stage renal disease with chronic dialysis not excluded)
* left ventricular ejection fraction <50% by echocardiography
* documented active malignancy
* chronic inflammatory disease
* planned coronary intervention or endovascular therapy or bypass surgery within 3 months
* known drug allergy history for cilostazol
* current use of cilostazol or any other cAMP-elevator
* premenopausal women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Circulating EPCs Number | 3 months
  Peripheral blood mononuclear cells (one million cells in each) are suspended in 100 µL phosphate-buffered saline and incubated for 30 min with monoclonal antibodies against human peridinin chlorophyll protein-conjugated cluster of differentiation antigen-45, phycoerythrin-conjugated anti-human cluster of differentiation antigen-34 antibody and anti-human kinase insert domain receptor (KDR) antibody conjugated with Alexa Flour 647. Cells are washed and analyzed on a FACSCalibur flow cytometer with 100,000 events in the lymphocyte gate. EPCs, which are defined as negative for cluster of differentiation antigen-45 and positive for cluster of differentiation antigen-34 and KDR. Based on the peripheral blood mononuclear cell counts, the absolute number of circulating EPCs/µL is calculated.

SECONDARY OUTCOMES:
Colony Formation by EPCs | 3 months
  Peripheral blood mononuclear cells are isolated by density gradient centrifugation according to standard protocols. After centrifugation, cells are washed, resuspended in M199 medium supplemented with 20% (vol/vol) fetal bovine serum, 10 ng/ml vascular endothelial growth factor, 2 ng/ml basic-fibroblast growth factor, 10 ng/ml epidermal growth factor and 2 ng/ml insulin growth factor, and cultured in 24-well plates coated with human fibronectin for 7 days. EPCs cells are confirmed by uptake of acetyl-low density lipoprotein and lectin and by the expression of EPC markers. Cells are harvested after 7 days, fixed and stained with crystal violet reagent. The colony densities are quantified with an Olympus microscope at 100-fold magnification using an imaging measurement software.

OTHER OUTCOMES:
Viability (Proliferation) of EPCs | 3 months
  250,000 cells are seeded in each well of a 96-well plate and the cells are added with 200 μl of the culture medium and incubated at 37°C. Medium change is performed 3 days later. On 7th day, the plate is then re-incubated with 100 μl fresh medium and additional 50 μl of 2,3-Bis-(2-Methoxy-4-Nitro-5-Sulfophenyl)-2 Hydrogen-Tetrazolium-5-Carboxanilide reagent, and further incubated in dark at 37°C for 4 h. After incubation, the orange colored complex formed is read at 450 nm using a microplate reader with a 450 nm reference filter.

CONTACTS AND LOCATIONS:
Overall Officials: Ting-Hsing Chao, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Background] Chao TH, Tseng SY, Li YH, Liu PY, Cho CL, Shi GY, Wu HL, Chen JH. A novel vasculo-angiogenic effect of cilostazol mediated by cross-talk between multiple signalling pathways including the ERK/p38 MAPK signalling transduction cascade. Clin Sci (Lond). 2012 Aug 1;123(3):147-59. doi: 10.1042/CS20110432. PMID 22339730
- [Background] Biscetti F, Pecorini G, Straface G, Arena V, Stigliano E, Rutella S, Locatelli F, Angelini F, Ghirlanda G, Flex A. Cilostazol promotes angiogenesis after peripheral ischemia through a VEGF-dependent mechanism. Int J Cardiol. 2013 Aug 10;167(3):910-6. doi: 10.1016/j.ijcard.2012.03.103. Epub 2012 Apr 2. PMID 22473072
- [Derived] Chao TH, Chen IC, Li YH, Lee PT, Tseng SY. Plasma Levels of Proprotein Convertase Subtilisin/Kexin Type 9 Are Elevated in Patients With Peripheral Artery Disease and Associated With Metabolic Disorders and Dysfunction in Circulating Progenitor Cells. J Am Heart Assoc. 2016 May 20;5(5):e003497. doi: 10.1161/JAHA.116.003497. PMID 27207972